CLINICAL TRIAL: NCT01987076
Title: DRESS - Setting of Corticosteroid Treatment.
Brief Title: Comparison Between Corticosteroid and Topical Steroids in the DRESS
Acronym: DRESSCODE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P110108; 2012-001471-36 (EudraCT Number)
Record Dates: First submitted 2013-09-17; First posted 2013-11-19 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Drug Rash With Eosinophilia and Systemic Symptoms
Keywords: DRESS; Systemic steroid; Topical steroid; Treatment
MeSH Terms: conditions — Drug Hypersensitivity Syndrome | interventions — Prednisone; Clobetasol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticosteroids per os: Prednisone + Emollient (Active Comparator)
  Interventions: Drug: Prednisone
- Topical corticosteroid: Clobetasol + Emollient (Experimental)
  Interventions: Drug: Clobetasol

INTERVENTIONS:
Drug: Prednisone — Prednisone:
  Day 0 to day 30: 0.5mg/kg/day Day 30 to day 180: doses decreasing from 15 to 25% every 15 days until Day75 and 10 to 15% every 15 days.
  Arms: Corticosteroids per os: Prednisone + Emollient
Drug: Clobetasol — Clobetasol: cream 0.05% Day 0 to day 30: 30 grams per day Day 30 to day 45: 20 grams per day Day 45 to day 60: 20 grams every other day Day 60 to day 120: 20 grams biweekly Day 120 to day 150: 20 grams one a week
  Arms: Topical corticosteroid: Clobetasol + Emollient

SUMMARY:
Drug reaction with eosinophilia and systemic symptoms (DRESS) is a rare and severe multiorgan adverse drug reaction occurring within 2 to 6-8 weeks after a new drug intake. DRESS syndrome is defined by the combination of clinical manifestations, cutaneous, visceral and biological disturbances. Its prognosis is directly linked to severity of visceral involvement, with a mortality evaluated above 10%.

Considering curative treatment, there is no consensus. Until now, no controlled trial has been performed. Systemic steroids are mainly used in first intention, in particular for management of visceral involvements, whatever their severity. From clinical practice, topical steroids are often used and could be helpful in the therapeutic management of DRESS.

We propose to evaluate systemic steroids versus very potent topical steroids in a multicentric randomized controlled trial including defined moderate DRESS, ie the non-inferiority of very potent topical steroids in terms of remission of visceral involvement at Day30 and the superiority of very potent topical steroids in terms of delay to remission of skin involvement.

ELIGIBILITY:
Inclusion Criteria:

* patient age ≥ 18 years
* signing informed consent form
* DRESS diagnosis with at least 4 criteria a, b, c, d

  1. Skin rash occurring at least 10 days and not more than two months after continuous drug intake (or within less than 10 days in case of rechallenge)
  2. Fever ≥ 38 ° at the time of examination or fever ≥ 38.5 ° peak in the last 72 hours (amendment 2 : ANSM + CPP : 08/04/14)
  3. at least one visceral compatible :
* lymphadenopathy on at least two different sites measuring at least 1 cm in diameter
* transaminases > 2 upper limit of normal (ULN) or alkaline phosphatise > 3 ULN
* lung involvement defined by hypoxemia (capillary oximetry ≤ 95%) and/or interstitial lung disease on chest radiography or scanner, in absence of other lung disease
* myocarditis, pericarditis (ECG clinical suspicion and confirmed by echocardiography)
* renal impairment defined as creatinine increase above the normal laboratory value associated with leucocyturia > 1000 / mm3 or proteinuria, a Na / K ratio >1 and Urine Cyto-bacteriology (EBCU) sterile in the absence of preexisting renal disease d) At least one of the following haematological abnormalities:
* eosinophilia ≥ 0.7 g/l or > 10 % absolute
* lymphocytosis ≥ 5*10^9 /l
* presence of atypical blood lymphocytes
* Patient with moderate DRESS : defined by at least one reached as follows :
* pulmonary: interstitial pneumonia with oxygen partial pressure in arterial blood (PaO2) 60-75 mmHg without dyspnoea at rest
* Hepatic: transaminases ≥ 4 ULN and < 15 ULN and/or PAL ≥5 ULN and V factor 50% (amendment 2 : ANSM + CPP : 08/04/14)
* renal :
* acute renal failure and organic sharp increase in the 48 hours preceding the inclusion of more of 26.4 micromol/l creatinine
* and / or increase of 1.5 times the normal creatinine value
* and / or decrease of oliguria of less than 0.5 ml/kg/h followed by a 6 hours
* cord: pancytopenia (7≤Hb≤10 gr/dl and/or 50<p<100 G/L, 0.5<PNN≤1.5G/l)
* AND absence of cardiac, neurological or gastrointestinal (gut, pancreas) threatening
* Drug withdrawal
* Patient with health insurance (or entitled beneficiary)
* Patient accepting the constraints of the test

Exclusion Criteria:

* uncontrolled sepsis
* unability to discontinue the medication(s) due
* known hypersensitivity to systemic or topical corticosteroids
* hepatitis B or C known, (active HIV status known suppressed by amendment 5 : ANSM16/04/2015 and CPP 07/04/2015)
* (Patient already treated by corticosteroid :

  * More than 48 hours
  * Less than 48 hours to following conditions :
* Patients receiving more than 1 mg/kg/day of prednisone per os
* Patients receiving methylprednisolone pulse up to 1mg/kg prednisone equivalent
* (Patients receiving more than 30 grams per day level 3 topical steroid or more than 10 grams per day level 4 topical steroid --> suppressed by amendment 3 : ANSM 28/05/14 CPP : 10/06/14)
* (Patient undergoing immunosuppressive therapy for another disease suppressed by amendment 5 : ANSM16/04/2015 and CPP 07/04/2015)
* Participation in another drug biomedical research
* Primitive bacterial infections, fungal or parasitic
* Severe rosacea cont-indicating the use of corticosteroid
* Presence of at least one ulcerated lesion (more than 10cm2)
* Severe dermatitis perioral cont-indicating the use of corticosteroid
* Severe acne contra-indicating the use of a corticosteroid
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Rate of patients with a complete or almost healing of visceral involvement to D30 +/- 5 days AND complete or almost complete healing of skin involvement. | Day 30

SECONDARY OUTCOMES:
Rate of patients with a complete or almost complete healing of cutaneous and visceral involvement at Day 30 ± 5 days | Day 30
Delays of complete or almost complete visceral healing | Month 12
Relapse rates and bounces rates between the end of acute treatment and M12 | Month 12
Patients rate evaluating to severe form (occurrence of a criterion defining the severe form cf. Above) | Month 12
Occurrence rate of moderate DRESS visceral involvement, during the initial treatment (D0 to D30) not existing at inclusion | Day 30
Mortality rate at Month 12 | Month 12
Sequelae rate at Month 12 | Month 12
Systemic steroids adverse reactions rate | Month 12
Topical steroids adverse reactions rate | Month 12
Patch tests evaluation in DRESS | Month 6
Reactivation kinetics of Cytomegalovirus (CMV), Epstein-Barr virus (EBV), Herpes Simplex virus (HSV), Human Herpes virus6 (HHV6) and Human Herpes virus7 (HHV7) | Day 0, Day 7, Day 14, Day 21, Day 30, Month 3, Month 6, Month 12
Predictive value of lymphocyte transformation test in imputability | Day 0, Day 30, Month 6, Month 12
Immunological factors evaluation in the skin | Day 30
Blood inflammatory cytokines and chemokines analysis | Day 0, Day 30, Month 6
Blood cytokines polymorphisms analysis | Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CHOSIDOW, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Eshki M, Allanore L, Musette P, Milpied B, Grange A, Guillaume JC, Chosidow O, Guillot I, Paradis V, Joly P, Crickx B, Ranger-Rogez S, Descamps V. Twelve-year analysis of severe cases of drug reaction with eosinophilia and systemic symptoms: a cause of unpredictable multiorgan failure. Arch Dermatol. 2009 Jan;145(1):67-72. doi: 10.1001/archderm.145.1.67. PMID 19153346
- [Background] Mardivirin L, Valeyrie-Allanore L, Branlant-Redon E, Beneton N, Jidar K, Barbaud A, Crickx B, Ranger-Rogez S, Descamps V. Amoxicillin-induced flare in patients with DRESS (Drug Reaction with Eosinophilia and Systemic Symptoms): report of seven cases and demonstration of a direct effect of amoxicillin on Human Herpesvirus 6 replication in vitro. Eur J Dermatol. 2010 Jan-Feb;20(1):68-73. doi: 10.1684/ejd.2010.0821. Epub 2009 Oct 12. PMID 19822481
- [Derived] Funck-Brentano E, Duong TA, Bouvresse S, Bagot M, Wolkenstein P, Roujeau JC, Chosidow O, Valeyrie-Allanore L. Therapeutic management of DRESS: a retrospective study of 38 cases. J Am Acad Dermatol. 2015 Feb;72(2):246-52. doi: 10.1016/j.jaad.2014.10.032. PMID 25592341